CLINICAL TRIAL: NCT00863473
Title: Health and Cost Consequenses of Surgical Versus Conservative Treatment for a Comminuted Humerus Fracture. Do Interlocking Plate Surgery Benefit Displaced Proximal Humerus Fractures? A Randomized Clinical Trial
Brief Title: Comminuted Proximal Humeral Fractures. A Randomised Study of Surgical Versus Conservative Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Aker (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Tore Fjalestad, MD PhD Consultant, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AkerU_s422
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Proximal Humeral Fracture; Osteosynthesis or Conservative Treatment
Keywords: Proximal Humerus Fracture in elderly
MeSH Terms: conditions — Shoulder Fractures | interventions — Surgical Procedures, Operative

ARMS (2):
- Conservative /Physiotherapy (No Intervention): Active training protocol with instructed physiotherapy and self excercises
- Surgery with LCP T plate (Active Comparator): Surgical treatment with interlocking plate
  Interventions: Procedure: Surgical treatment with LCP

INTERVENTIONS:
Procedure: Surgical treatment with LCP
  Arms: Surgery with LCP T plate

SUMMARY:
1. Do a standardized surgical treatment of unstable displaced proximal humerus fracture in patients aged over 60 compared to a standardized conservative treatment gain a better functional outcome after one year?
2. Do surgical treatment gain more QALY than conservative treatment after one year?

ELIGIBILITY:
Inclusion Criteria:

* proximal humerus fracture of AO group B2 or C2 (displaced fracture of extra-articular or articular, bifocal type) admitted in hospital

Exclusion Criteria:

* aged less than 60 year
* patients of non-Scandinavian ethnicity
* previous history of injury or illness of the injured or contralateral shoulder
* injury of other part of the humerus or the contralateral upper extremity,
* alcohol- or drug abuse
* dementia or neurological diseases
* severe cardiovascular disease that would contraindicate surgery

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Functional shoulder score according to Constant (Original described Differences between the injured and uninjured shoulder as well as Adjusted according to age and gender). | 12 and 24 months

SECONDARY OUTCOMES:
QALY (HRQoL score according to Harri Sintonen 15D and Costs) | 12 and 24 months
ASES score (modified self assessment) C) Radiographic score | 12 and 24 months
Radiographic score | 12 and 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tore Fjalestad, Ortopeadic Dept, Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Background] Fjalestad T, Hole MO, Hovden IA, Blucher J, Stromsoe K. Surgical treatment with an angular stable plate for complex displaced proximal humeral fractures in elderly patients: a randomized controlled trial. J Orthop Trauma. 2012 Feb;26(2):98-106. doi: 10.1097/BOT.0b013e31821c2e15. PMID 21804410
- [Background] Fjalestad T, Hole MO, Jorgensen JJ, Stromsoe K, Kristiansen IS. Health and cost consequences of surgical versus conservative treatment for a comminuted proximal humeral fracture in elderly patients. Injury. 2010 Jun;41(6):599-605. doi: 10.1016/j.injury.2009.10.056. Epub 2009 Nov 27. PMID 19945102
- [Background] Fjalestad T, Hole MO. Displaced proximal humeral fractures: operative versus non-operative treatment--a 2-year extension of a randomized controlled trial. Eur J Orthop Surg Traumatol. 2014 Oct;24(7):1067-73. doi: 10.1007/s00590-013-1403-y. Epub 2014 Jan 11. PMID 24413845